CLINICAL TRIAL: NCT03081039
Title: A Phase III, Multicenter, Open-Label, Randomized Study of Cisplatin or Carboplatin With Gemcitabine Versus Gemcitabine Alone as Adjuvant Therapy in Patients With Resected or Ablated Intra-Hepatic Cholangiocarcinoma
Brief Title: A Study of Cisplatin or Carboplatin With Gemcitabine Versus Gemcitabine Alone as Adjuvant Therapy in Patients With Resected or Ablation Intra-Hepatic Cholangiocarcinoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Competing study
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Robert C. Martin, Principal Investigator, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UL 2016.1
Record Dates: First submitted 2017-02-09; First posted 2017-03-15 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2017-03

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: cholangiocarcinoma; gemcitabine; carboplatin; cisplatin
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Carboplatin; Cisplatin; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to one of two treatment arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Cisplatin or Carboplatin with Gemcitabine for 6 cycles
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Gemcitabine
- Arm B (Active Comparator): Gemcitabine alone for 6 cycles
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Carboplatin — Arm A: Carboplatin or Cisplatin every 21 days for 6 cycles. Dose based on weight.
  Arms: Arm A
Drug: Cisplatin — Arm A: Cisplatin or Carboplatin every 21 days for 6 cycles. Dose based on weight.
  Arms: Arm A
Drug: Gemcitabine — Arm A: Given with either Cisplatin or Carboplatin every 21 days for 6 weeks. Dose based on individuals weight.
  Arm B: Gemcitabine alone every 21 days for 6 cycles. Dose based on weight.

SUMMARY:
Compare the efficacy of adjuvant chemotherapy with Cisplatin or Carboplatin and Gemcitabine versus Gemcitabine in patients with resected or ablated intra-hepatic cholangiocarcinoma.

DETAILED DESCRIPTION:
Phase III, multicenter, open label, randomized study of Cisplatin or Carboplatin with Gemcitabine versus Gemcitabine alone as adjuvant therapy in patients with resected or ablated intra-hepatic cholangiocarcinoma. Subjects will be randomized in a 1:1 fashion to Cisplatin or Carboplatin with Gemcitabine versus Gemcitabine alone.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, of any race or sex who are eligible to sign written consent and have undergone prior resection of histological evidence of intrahepatic cholangiocarcinoma
* Hematologic function: ANC ≥ 1.5 x 10 /L, platelets ≥ 75 x 10 /L, and hemoglobin > 9 g/dL
* Adequate liver function as measured by: total bilirubin ≤ 2.0 mg/dl, AST and ALT ≤ 5 ULN, albumin ≥ 2.5 g/dl
* Adequate renal function as measured by: creatinine ≤ 2.9 mg/dl, > 50 ml/min calculated by the C-G equation
* Non-pregnant women of child bearing potential and fertile men are required to use effective contraception (negative pregnancy test for women of child-bearing age)
* ECOG status ≤ 1 at screening

Exclusion Criteria:

* Subjects will be eligible for the study if they meet all inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2022-04-28 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Every three months for 4 years

SECONDARY OUTCOMES:
Progression Free Survival | Every three months for 4 years.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Martin, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No